CLINICAL TRIAL: NCT03615040
Title: A Randomised Placebo-controlled Trial of Anti-ST2 in COPD (COPD-ST2OP)
Brief Title: Anti-ST2 (MSTT1041A) in COPD (COPD-ST2OP)
Acronym: COPD-ST2OP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Glenfield Hospital, Leicester (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0671; 2018-000919-24 (EudraCT Number); GB40568 (Other Grant/Funding Number: Genentech); U1111-1210-1335 (Other: WHO Universal Trial Number); 244758 (Other: IRAS Number); 18/EM/0189 (Other: East Midlands - Leicester South Research Ethics Committee)
Record Dates: First submitted 2018-05-04; First posted 2018-08-03 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2020-06

CONDITIONS: COPD Exacerbation
Keywords: COPD; Exacerbations; ST2 MAb; RG6149; MSTT1041A; Anti-ST2; Phase IIa; Placebo controlled
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — astegolimab

STUDY DESIGN:
Intervention Model Description: Single-centre, double-blinded, placebo-controlled, parallel group, randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A or B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anti-ST2 (Experimental): Anti-ST2 (MSTT1041A) received as subcutaneous injection by infusion pump at 490mg every 4 weeks over a 48 week treatment period.
  Interventions: Drug: MSTT1041A
- Placebo (Placebo Comparator): Placebo (no active component) received as subcutaneous injection by infusion pump at 490mg every 4 weeks over a 48 week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSTT1041A — MSTT1041A (RO7187807; formerly made by Amgen [AMG] and referred to as AMG 282) is a novel biopharmaceutical that blocks signaling of interleukin (IL)-33, an inflammatory cytokine of the IL-1 family and member of the newly discovered "alarmin" class of molecules. IL-33 is released from airway epithelial cells in response to allergens, irritants, and infection. IL-33 release can trigger acute exacerbations in both asthma and COPD. MSTT1041A has the ability to block inflammation,prevent exacerbations, and improve lung function and quality of life.
  Anti-ST2 is presented as sterile, clear, and colourless to slightly yellow liquid. Each sterile vial is filled with a 1 mL deliverable volume of 70 mg/mL. It is formulated with 15 mM sodium acetate, 9.0% (w/v) sucrose, 0.01% (w/v) polysorbate 20, pH 5.2.
  Other Names: RO7187807; ST2 MAb; Anti-ST2; AMG 282; RG6149
  Arms: Anti-ST2
Drug: Placebo — Placebo for Anti-ST2 (MSTT1041A) is formulated with 10 mM sodium acetate, 9.0% (w/v) sucrose, 0.004% (w/v) polysorbate 20, pH 5.2, and is supplied in an identical vial configuration.
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a significant cause of morbidity and mortality worldwide. In contrast to other chronic diseases, COPD is increasing in prevalence and is projected to be the third-leading cause of death and disability worldwide by 2030. The costs to society for treating COPD are high, accounting for approximately 3.4% of the total health care budget of the European Union. Acute exacerbations of COPD (AECOPD) are responsible for a large portion of the economic burden of COPD. More than 500,000 hospitalisations and 100,000 deaths are attributed to AECOPD in the US each year. In addition to a substantial economic burden, AECOPD is also responsible for much of the morbidity and mortality from COPD.

Interleukin-33 (IL-33) is an alarmin released from the epithelium following damage. IL-33 is an IL-1 family alarmin cytokine constitutively expressed at epithelial barrier surfaces where it is rapidly released from cells during tissue injury. IL-33 signals through a receptor complex of IL-1 receptor-like 1 (IL1RL1) (known as ST2) and IL-1 receptor accessory protein (IL1RAcP) to initiate MyD88-dependent inflammatory pathways. The role of the IL33/ST2 axis in COPD is uncertain. IL33 has been implicated in eosinophil recruitment to the airway and maturation in the bone marrow largely via its effects upon innate lymphoid cells. IL33 increased following experimental cold in asthma and thus might play a role in the consequent inflammatory response and possible susceptibility to secondary bacterial infection in obstructive lung disease. Both eosinophilic inflammation and viral infection drive COPD exacerbations and therefore targeting the IL33/ST2 axis might reduce COPD exacerbations.

The main aim of this trial is to evaluate whether anti-ST2 will impact on airway inflammation in COPD and therefore reduce the frequency of exacerbations. For the purposes of this trial, exacerbations are defined as flare-ups of symptoms involving the use of healthcare resulting in treatment with steroids and/or antibiotics and/or hospitalisation or death due to COPD.

DETAILED DESCRIPTION:
This is a single-centre, double-blind, placebo- controlled, parallel group, randomised controlled trial to assess the efficacy and safety of anti-ST2 compared to placebo, in patients with moderate to very severe COPD (GOLD II-IV). Anti-ST2 will be administered via subcutaneous injection once every 4 weeks (Week 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44) during the 48-week treatment period. Participants will be followed up for 60 weeks (i.e. 48 week treatment period and 12 week follow-up), with secondary outcome measures at baseline, 4, 12, 24, 36, 48 and 60 weeks and at exacerbation events presenting prior to treatment initiation.

After signing the informed consent at the initial visit, patients will enter a screening period which should last for up to 2 weeks unless extension of the screening period is necessary under certain circumstances. Patients who qualify to participate in the study will be randomised into a 48-week treatment period in which they will receive either 490 mg anti-ST2 or a matching placebo. Patients will be evaluated for an additional 12 weeks following completion of the randomised treatment period. Treatment groups will remain blinded until the 60-week follow-up period is completed, and trial database is locked.

This trial is sponsored by the University of Leicester, coordinated by the National Institute for Health Research (NIHR) Biomedical Research Centre (BRC) - Respiratory and Leicester Clinical Trials Unit (LCTU) and funded by Genentech, Inc.

The primary objective of the study is to evaluate the efficacy of anti-ST2 versus placebo on frequency of moderate-to-severe exacerbations (health care utilisation resulting in treatment with systemic corticosteroids and/or antibiotics or hospitalisation, respectively) as add-on to standard of care.

Secondary objectives: another key objective is to assess the safety and tolerability of subcutaneous (SC) doses of anti-ST2 compared to placebo in adult patients with moderate to very severe COPD.

Additionally, to assess the effects of anti-ST2 versus placebo both during stable visits and at the exacerbation events on the following:

1. Symptoms
2. Health status
3. Lung function
4. Inflammatory cell differentials i. Sputum cell count ii. Blood cell count
5. Airway morphometry
6. Pharmacogenomics

Exploratory objectives include:

1. Systemic inflammation
2. Upper airway inflammation
3. Airway infection and ecology
4. Breath volatile organic compound profiling
5. Quantitative airway geometry and densitometry
6. Pharmacogenomics
7. Pharmacokinetics and ADA level
8. Pharmacogenomics response analysis in subgroups determined by SNPs for alleles associated with the IL33/ST2 axis.

Subgroup objectives: to evaluate the efficacy of anti-ST2 versus placebo on the outcome rate of protocol-defined COPD exacerbations through 48 weeks treatment period, patient reported outcomes (PROs) [SGRQ-c], and lung function [FEV1] in subgroups defined by baseline blood eosinophil count.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms typical of COPD when stable (baseline mMRC dyspnoea score ≥ 2)
2. GOLD COPD stage 2-4
3. Smoking pack years ≥ 10 years
4. Age > 40 years
5. Receiving standard-of-care drug therapy as per British Thoracic Society (BTS) guidance for COPD
6. A history of ≥ 2 moderate-to-severe exacerbations in the last 12 months.
7. Be able to give valid written consent; compliant with study procedures and study visits.
8. Able to understand written and spoken English

Exclusion Criteria:

1. Significant known respiratory disorders other than COPD that in the view of the investigator will affect the study
2. Patients whose treatment is considered palliative (life expectancy <12 months)
3. Known hypersensitivity to the active substance of the investigational product (IP) or any of the excipients
4. Known history of anaphylaxis
5. Patients with a COPD exacerbation and/or pneumonia within the 4 weeks prior to visit 1
6. Have, in the opinion of investigator, uncontrolled co-morbid conditions, such as diabetes mellitus, hypertension and heart failure [e.g. New York Heart Association (NYHA) class III (e.g. less than ordinary activity causes fatigue, palpitation, or dyspnoea), and class IV (e.g. Symptoms of heart failure at rest)] that will affect the study.
7. Myocardial infarction, unstable angina or stroke within 12 month prior to screening
8. Diagnosis of malignancy within 5 years of visit 1 (except for excised localised carcinoma of skin not including malignant melanoma)
9. Clinically significant ECG changes, which in the opinion of investigator warrants further investigations
10. Laboratory abnormalities, which in the opinion of investigator warrants further investigations
11. Have, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse.
12. Pregnant, breastfeeding, or lactating women. Women of child-bearing potential (i.e. not surgically sterilised or post- menopausal) must have a negative blood serum pregnancy test performed at the screening visit and must agree to use two methods of birth control, (one of which must be a barrier method).
13. Participation in an interventional clinical study within 3 months of visit 1 or receipt of any investigational medicinal product within 3 months or 5 half- lives.
14. Upon questioning the patient has blood born infection (e.g. HIV, hepatitis B or C)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brightling, Prof, Principal Investigator — University of Leicester
Locations (1):
- Biomedical Research Centre- Respiratory, Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yousuf AJ, Mohammed S, Carr L, Yavari Ramsheh M, Micieli C, Mistry V, Haldar K, Wright A, Novotny P, Parker S, Glover S, Finch J, Quann N, Brookes CL, Hobson R, Ibrahim W, Russell RJ, John C, Grimbaldeston MA, Choy DF, Cheung D, Steiner M, Greening NJ, Brightling CE. Astegolimab, an anti-ST2, in chronic obstructive pulmonary disease (COPD-ST2OP): a phase 2a, placebo-controlled trial. Lancet Respir Med. 2022 May;10(5):469-477. doi: 10.1016/S2213-2600(21)00556-7. Epub 2022 Mar 24. PMID 35339234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at a single centre. Potential participants were identified by the research team using a variety of methods: database of previous COPD trial participants who consented to be contacted for future trials; respiratory outpatient clinics/acute admission unit; self-referrals; GP practices. Recruitment ran between 11 Oct 2018 and 05 Jul 2019.
Pre-assignment Details: Potential participants were assessed according to eligibility criteria at initial screening and provided written informed consent before commencing any trial-related procedures. Participants then entered a screening period for 7-14 days before randomisation. eligible to participate were randomised into a 48-week treatment period (anti-ST2/placebo).
Groups:
- Anti-ST2: Anti-ST2 (MSTT1041A*) received as subcutaneous injection by infusion pump at 490mg every 4 weeks over a 48 week treatment period.
  Anti-ST2 was presented as sterile, clear, and colourless to slightly yellow liquid. Each sterile vial is filled with a 1 mL deliverable volume of 70 mg/mL. It was formulated with 15 mM sodium acetate, 9.0% (w/v) sucrose, 0.01% (w/v) polysorbate 20, pH 5.2.
  *Official USAN name for MSTT1041A is now astegolimab
- Placebo: Placebo (no active component) received as subcutaneous injection by infusion pump at 490mg every 4 weeks over a 48 week treatment period.
  Placebo for Anti-ST2 (MSTT1041A) was formulated with 10 mM sodium acetate, 9.0% (w/v) sucrose, 0.004% (w/v) polysorbate 20, pH 5.2, and was supplied in an identical vial configuration.
Period: Overall Study
Arm/Group | Anti-ST2 | Placebo
Started | 42 | 39
Completed | 36 | 34
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Clinical diagnosis of lung cancer | 1 | 0
Not completed — Clinical diagnosis of oesophageal cancer | 1 | 0
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-ST2 | Placebo | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 30 | 35 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.2) | 70.8 (6.2) | 69.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 25 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 39 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 39 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Moderate to Severe Exacerbation (Defined as Requiring Treatment With Systemic Corticosteroids and/or Antibiotics in the Community or Hospital or Hospitalisation).
Description: Where a COPD exacerbation is defined by symptomatic worsening of COPD requiring:
  * Use of systemic corticosteroids for at least 3 days; a single depot injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids; and/or
  * Use of antibiotics and/or
  * inpatient hospitalisation or death due to COPD
Time Frame: 0-48 weeks
Population: An intention-to-treat population was used for the primary analysis and all participants were included in the analysis (n = 81). The primary analysis used observed data, meaning only observed exacerbations were used alongside the corresponding time period in the offset of log-time.
Measure: Mean (Standard Deviation); unit: Exacerbations
Groups:
- Anti-ST2: Anti-ST2 (MSTT1041A) received as subcutaneous injection by infusion pump at 490mg every 4 weeks over a 48 week treatment period.
  MSTT1041A: MSTT1041A (RO7187807; formerly made by Amgen [AMG] and referred to as AMG 282) is a novel biopharmaceutical that blocks signaling of interleukin (IL)-33, an inflammatory cytokine of the IL-1 family and member of the newly discovered "alarmin" class of molecules. IL-33 is released from airway epithelial cells in response to allergens, irritants, and infection. IL-33 release can trigger acute exacerbations in both asthma and COPD. MSTT1041A has the ability to block inflammation,prevent exacerbations, and improve lung function and quality of life.
  Anti-ST2 is presented as sterile, clear, and colourless to slightly yellow liquid. Each sterile vial is filled with a 1 mL deliverable volume of 70 mg/mL. It is formulated with 15 mM sodium acetate, 9.0% (w/v) sucrose, 0.01% (w/v) polysorbate 20, pH 5.2.
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
Exacerbations | 2.21 (2.04) | 2.67 (2.14)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; A generalised linear model (assuming neg. binomial distribution) was used. The model includes the number of exacerbations during the 48 week treatment as an outcome with explanatory variables of treatment arm & number of exacerbations in the 12 months prior to the trial (stratification factor), and log-time on trial (in weeks) as an offset. The offset, allows for different lengths of time in the trial. Only observed exacerbations were used alongside the corresponding time period in the offset; Test type: Superiority; p = 0.195, t-test, 2 sided; Incidence Rate Ratio = 0.78, 95% CI 2-sided [0.53 to 1.14], Standard Error of Mean 0.15

2. Secondary Outcome: Adverse Event Rate in the 48 Weeks of the Trial From First Dose
Description: Number of Participants with Adverse Events in the 48 Weeks of the Trial From First Dose
Time Frame: Weeks 0 , 4, 12, 24, 26, 48
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
Participants | 34 | 28

3. Secondary Outcome: Serious Adverse Event Rate in the 48 Weeks of the Trial From First Dose
Description: Number of Participants with Serious Adverse Events in the 48 Weeks of the Trial From First Dose
Time Frame: Weeks 0 , 4, 12, 24, 26, 48
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
Participants | 12 | 16

4. Secondary Outcome: St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Total Score
Description: Patient reported outcome (PRO). To evaluate health status; designed to measure health impairment in patients with asthma and COPD. It is in two parts. Part I produces the Symptoms score, and Part 2 the Activity and Impact scores. A Total score is also produced. The Total score is calculated by summing the weights to all the positive responses in each component. This score is then put onto the scale 0 to 100 by dividing by the Total possible sum (3201.9)- and times by 100. A score of 0 would represent the best health and a score of 100 would represent the worst possible state of the patient.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
score on a scale
  Baseline | 60.1 (13.7) | 58.4 (17.6)
  Week 4: number analyzed (Participants) | 42 | 38
  Week 4 | 56.7 (13.5) | 58.9 (16.5)
  Week 12: number analyzed (Participants) | 42 | 35
  Week 12 | 56.9 (15.2) | 59.9 (18.2)
  Week 24: number analyzed (Participants) | 40 | 36
  Week 24 | 56.6 (15.3) | 59.6 (17.9)
  Week 36: number analyzed (Participants) | 39 | 35
  Week 36 | 59.5 (14.6) | 59.5 (17.0)
  Week 48: number analyzed (Participants) | 20 | 16
  Week 48 | 57.7 (15.7) | 63.3 (17.2)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Calculated using mixed effect linear model with dependent variable of the outcome at baseline and follow-up time points (Week 4, 12, 24, 36, 48); explanatory variables of treatment arm, number of exacerbations in the 12 months prior to the trial (stratification factor), visit time point (as categorical variable), baseline score; an interaction term between treatment and visit as fixed effects; and patient identification as a random effect; Test type: Superiority; p = 0.039, Mixed Models Analysis; Mean Difference (Net) = -3.3, 95% CI 2-sided [-6.4 to -0.2]

5. Secondary Outcome: COPD Assessment Test (CAT) (Questionnaire)
Description: Patient reported outcome (PRO). To evaluate health status: evaluation and rehabilitation education guidance on the respiratory and motor functions of patients with chronic obstructive pulmonary disease. CAT score is made by summing the score to eight questions on COPD. For each, the person with COPD picks the number between 0-5 that reflects their response. A zero indicates no effect on quality of life, whereas a 5 suggests a very significant effect.The CAT has a scoring range of 0-40, with 40 indicating the most severe COPD and 0 being the least severe COPD.
  A change of 2 units suggests a meaningful difference. This test should be used in conjunction with the mMRC and forced expiratory volume in one second (FEV1) to determine COPD health assessment of participants.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
score on a scale
  Week 0 | 22.1 (6.6) | 22.6 (5.7)
  Week 4: number analyzed (Participants) | 42 | 38
  Week 4 | 22.2 (5.5) | 21.7 (5.8)
  Week 12 | 22.0 (5.1) | 22.3 (6.9)
  Week 24: number analyzed (Participants) | 40 | 36
  Week 24 | 22.7 (6.9) | 22.1 (5.5)
  Week 36: number analyzed (Participants) | 39 | 35
  Week 36 | 22.7 (5.0) | 22.4 (6.0)
  Week 48: number analyzed (Participants) | 20 | 16
  Week 48 | 23.4 (6.0) | 23.6 (7.8)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.469, Mixed Models Analysis; Mean Difference (Net) = 0.53, 95% CI 2-sided [-0.91 to 2.00]

6. Secondary Outcome: Modified Medical Research Council (mMRC) Dyspnea Scale
Description: Patient reported outcome (PRO). To evaluate respiratory breathlessness symptoms (Grade 0-4, with Grade 0 being breathlessness with strenuous exercise to Grade 4 being breathlessness for daily activities like dressing).
Time Frame: Screening, weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
score on a scale
  Week 0 | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Week 4: number analyzed (Participants) | 42 | 38
  Week 4 | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Week 12: number analyzed (Participants) | 42 | 36
  Week 12 | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Week 24: number analyzed (Participants) | 40 | 36
  Week 24 | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0]
  Week 36: number analyzed (Participants) | 39 | 35
  Week 36 | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]
  Week 48: number analyzed (Participants) | 20 | 16
  Week 48 | 2.0 [2.0 to 3.0] | 2.0 [1.5 to 3.5]
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Wilcoxon Rank sum test of mMRC dyspnoea Week 4; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; Wilcoxon Rank sum test of mMRC dyspnoea Week 12; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Anti-ST2 vs Placebo; Wilcoxon Rank sum test of mMRC dyspnoea Week 24; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Anti-ST2 vs Placebo; Wilcoxon Rank sum test of mMRC dyspnoea Week 36; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Anti-ST2 vs Placebo; Wilcoxon Rank sum test of mMRC dyspnoea Week 48; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Visual Analogue Score (VAS) Total and Individual Dyspnoea, Cough, Sputum Production (100mm) Scores
Description: Patient reported outcome (PRO). To evaluate respiratory symptoms. The participant is asked to place a mark (X) on the scale at the point that best describes their health currently. Minimum score 0mm (better outcome), maximum score 100mm (worse outcome) for each section of the scale (dyspnoea, cough, sputum). The Total VAS score is the sum of the 3 scales, thus the minimum score is 0 (best outcome) and the maximum 300 (worst outcome).
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
units on a scale
  VAS Total Week 0 | 142.7 (54.6) | 143.8 (53.8)
  VAS Total Week 4: number analyzed (Participants) | 42 | 38
  VAS Total Week 4 | 129.3 (45.7) | 148.5 (61.2)
  VAS Total Week 12: number analyzed (Participants) | 42 | 35
  VAS Total Week 12 | 139.5 (50.3) | 140.0 (65.1)
  VAS Total Week 24: number analyzed (Participants) | 40 | 36
  VAS Total Week 24 | 131.0 (57.9) | 146.6 (55.1)
  VAS Total Week 36: number analyzed (Participants) | 39 | 20
  VAS Total Week 36 | 146.9 (51.9) | 147.6 (59.6)
  VAS Total Week 48: number analyzed (Participants) | 20 | 16
  VAS Total Week 48 | 140.7 (58.0) | 146.5 (70.0)
  VAS Dyspnoea Week 0 | 52.5 (20.3) | 53.5 (22.1)
  VAS Dyspnoea Week 4: number analyzed (Participants) | 42 | 38
  VAS Dyspnoea Week 4 | 50.1 (17.7) | 57.8 (20.6)
  VAS Dyspnoea Week 12: number analyzed (Participants) | 42 | 35
  VAS Dyspnoea Week 12 | 55.2 (17.1) | 54.7 (25.4)
  VAS Dyspnoea Week 24: number analyzed (Participants) | 40 | 36
  VAS Dyspnoea Week 24 | 46.5 (20.0) | 57.9 (22.6)
  VAS Dyspnoea Week 36: number analyzed (Participants) | 39 | 35
  VAS Dyspnoea Week 36 | 56.0 (18.6) | 57.6 (22.5)
  VAS Dyspnoea Week 48: number analyzed (Participants) | 20 | 16
  VAS Dyspnoea Week 48 | 58.8 (15.8) | 60.5 (21.8)
  VAS Cough Week 0 | 49.7 (23.7) | 47.5 (22.7)
  VAS Cough Week 4: number analyzed (Participants) | 42 | 38
  VAS Cough Week 4 | 41.3 (19.6) | 45.9 (25.5)
  VAS Cough Week 12: number analyzed (Participants) | 42 | 36
  VAS Cough Week 12 | 44.2 (22.3) | 45.1 (24.6)
  VAS Cough Week 24: number analyzed (Participants) | 40 | 35
  VAS Cough Week 24 | 47.6 (23.7) | 45.2 (21.9)
  VAS Cough Week 36: number analyzed (Participants) | 39 | 35
  VAS Cough Week 36 | 48.4 (20.4) | 46.0 (25.1)
  VAS Cough Week 48: number analyzed (Participants) | 20 | 16
  VAS Cough Week 48 | 40.4 (24.7) | 47.0 (29.6)
  VAS Sputum production Week 0 | 40.5 (25.5) | 42.8 (24.5)
  VAS Sputum production Week 4: number analyzed (Participants) | 42 | 38
  VAS Sputum production Week 4 | 37.9 (24.5) | 44.7 (27.0)
  VAS Sputum production Week 12: number analyzed (Participants) | 42 | 35
  VAS Sputum production Week 12 | 40.1 (25.7) | 40.2 (28.7)
  VAS Sputum production Week 24: number analyzed (Participants) | 40 | 36
  VAS Sputum production Week 24 | 36.9 (26.3) | 43.5 (24.3)
  VAS Sputum production Week 36: number analyzed (Participants) | 39 | 35
  VAS Sputum production Week 36 | 42.6 (27.3) | 44.0 (26.2)
  VAS Sputum production Week 48: number analyzed (Participants) | 20 | 16
  VAS Sputum production Week 48 | 41.5 (26.5) | 39.0 (27.6)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; VAS total; Test type: Superiority; p = 0.236, Mixed Models Analysis — Using mixed effect linear model with explanatory variables treatment, number of exacerbations in the 12 months prior to the trial (stratification), visit time point (as categorical variable) and baseline score as fixed effects; Mean Difference (Net) = -9.4, 95% CI 2-sided [-24.9 to 6.2]
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; VAS Dyspnoea; Test type: Superiority; p = 0.083, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -4.9, 95% CI 2-sided [-10.6 to 0.7]
Statistical Analysis 3: Comparison: Anti-ST2 vs Placebo; VAS Cough; Test type: Superiority; p = 0.546, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -2.1, 95% CI 2-sided [-8.9 to 4.7]
Statistical Analysis 4: Comparison: Anti-ST2 vs Placebo; VAS Sputum production; Test type: Superiority; p = 0.527, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -1.9, 95% CI 2-sided [-7.8 to 4.0]

8. Secondary Outcome: Sputum Purulence Colour Card
Description: The sputum purulence colour card using the Bronko test has values of 0, 1, 2, 3, 4, 5 and 6. Lower scores indicate better health.
Time Frame: Screening, week 12, 28, 36, 48
Population: Modified ITT (available data)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
score on a scale
  Week 0 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Week 12: number analyzed (Participants) | 42 | 36
  Week 12 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Week 24: number analyzed (Participants) | 40 | 36
  Week 24 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Week 36: number analyzed (Participants) | 38 | 36
  Week 36 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.5]
  Week 48: number analyzed (Participants) | 24 | 21
  Week 48 | 4.0 [2.0 to 6.0] | 4.0 [2.0 to 6.0]
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; sputum purulence colour card Week 12; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; sputum purulence colour card Week 24; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Anti-ST2 vs Placebo; sputum purulence colour card Week 36; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Anti-ST2 vs Placebo; sputum purulence colour card Week 48; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Pre and Post Bronchodilator (BD) Spirometry - FEV1/FVC Ratio
Description: To assess lung function. The participant will take a maximum inhalation, release maximum exhalation and then continue to exhale afterwards. They will then be treated with a bronchodilator. The spirometry test is then repeated to determine how much the bronchodilator medication helped with breathing. FEV1/FVC ratio will be calculated.
Time Frame: Week 0 and Week 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 8 | 5
Ratio
  Pre BD FEV1/FVC ratio Week 0 | 49.0 (14.1) | 46.6 (18.6)
  Pre BD FEV1/FVC ratio Week 48 | 51.0 (15.5) | 40.2 (9.6)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Pre BD FEV1/FVC ratio: Analysis of covariance (ANCOVA) adjusting for the baseline value; Test type: Superiority; p = 0.069, ANCOVA; Mean Difference (Final Values) = 9.06, 95% CI 2-sided [-0.83 to 18.97]

10. Secondary Outcome: Post BD Forced Expiratory Volume in 1 Second (FEV1)
Description: To assess lung function. FEV1 is the volume of air that can forcibly be blown out in first 1 second, after full inspiration. Post BD Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Screening, Weeks 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
Litres
  Week 0 | 1.21 (0.46) | 1.14 (0.48)
  Week 4: number analyzed (Participants) | 42 | 38
  Week 4 | 1.21 (0.46) | 1.09 (0.46)
  Week 12: number analyzed (Participants) | 42 | 34
  Week 12 | 1.22 (0.48) | 1.14 (0.52)
  Week 24: number analyzed (Participants) | 37 | 35
  Week 24 | 1.17 (0.43) | 1.10 (0.50)
  Week 36: number analyzed (Participants) | 37 | 33
  Week 36 | 1.23 (0.47) | 1.09 (0.52)
  Week 48: number analyzed (Participants) | 15 | 13
  Week 48 | 1.30 (0.50) | 1.09 (0.57)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; mixed effect linear model with explanatory variables of treatment arm, number of exacerbations in the 12 months prior to the trial (stratification factor), visit time point (as categorical variable), baseline score and patient identification as a random effect to account for repeated measures over time was fitted for each outcome. Adjusted mean difference between treatment arms with 95% confidence interval and p-value were reported. In the modified ITT population; Test type: Superiority; p = 0.094, Mixed Models Analysis; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.01 to 0.09]

11. Secondary Outcome: Body Plethysmography ('Body Box') Total Lung Capacity and Residual Volume
Description: To assess lung function, i.e. the functional residual capacity of the lungs. The participant sits inside an airtight box, inhales or exhales to a particular volume (usually FRC), and then a shutter drops across their breathing tube. The participant makes respiratory efforts against the closed shutter, causing their chest volume to expand and decompressing the air in their lungs. The increase in their chest volume slightly reduces the box volume (the non-person volume of the box) and thus slightly increases the pressure in the box. Total Lung Capacity and Residual Volume measured.
Time Frame: Week 0 and week 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 19 | 16
Litres
  Total Lung Capacity Week 0 | 7.5 (1.6) | 7.5 (1.4)
  Total Lung Capacity Week 48 | 7.6 (1.5) | 7.6 (1.5)
  Residual Volume Week 0 | 4.5 (1.5) | 4.7 (1.5)
  Residual Volume Week 48 | 4.8 (1.6) | 5.0 (1.4)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Total Lung Capacity; Test type: Superiority; p = 0.905, ANCOVA — To compare change from baseline to 48 weeks (pre and post treatment measurements), analysis of covariance (ANCOVA) model with baseline value as a covariate was fitted. Adjusted mean difference with 95% confidence interval and p-value were reported; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.46 to 0.52]
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; Residual Volume; Test type: Superiority; p = 0.775, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.62 to 0.47]

12. Secondary Outcome: Blood Inflammatory Cell Differentials
Description: To assess inflammation at exacerbation events. White blood cells, eosinophils and neutrophils will be measured.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Geometric Mean (Standard Error); unit: 10^9 *cells* per litre
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 42 | 39
10^9 *cells* per litre
  White Blood Cell Count Week 0 | 8.2 (0.045) | 8.0 (0.046)
  White Blood Cell Count Week 4: number analyzed (Participants) | 42 | 37
  White Blood Cell Count Week 4 | 7.5 (0.035) | 7.5 (0.037)
  White Blood Cell Count Week 12: number analyzed (Participants) | 42 | 35
  White Blood Cell Count Week 12 | 8.0 (0.043) | 7.7 (0.047)
  White Blood Cell Count Week 24: number analyzed (Participants) | 40 | 36
  White Blood Cell Count Week 24 | 7.8 (0.047) | 7.6 (0.050)
  White Blood Cell Count Week 36: number analyzed (Participants) | 39 | 36
  White Blood Cell Count Week 36 | 8.0 (0.046) | 7.3 (0.048)
  White Blood Cell Count Week 48: number analyzed (Participants) | 20 | 16
  White Blood Cell Count Week 48 | 7.5 (0.058) | 8.0 (0.065)
  Eosinophil Count Week 0 | 0.21 (0.107) | 0.20 (0.111)
  Eosinophil Count Week 4: number analyzed (Participants) | 42 | 37
  Eosinophil Count Week 4 | 0.15 (0.105) | 0.22 (0.111)
  Eosinophil Count Week 12: number analyzed (Participants) | 42 | 35
  Eosinophil Count Week 12 | 0.13 (0.105) | 0.20 (0.116)
  Eosinophil Count week 24: number analyzed (Participants) | 38 | 36
  Eosinophil Count week 24 | 0.12 (0.096) | 0.21 (0.099)
  Eosinophil Count Week 36: number analyzed (Participants) | 39 | 36
  Eosinophil Count Week 36 | 0.11 (0.106) | 0.20 (0.111)
  Eosinophil Count week 48: number analyzed (Participants) | 20 | 16
  Eosinophil Count week 48 | 0.10 (0.143) | 0.17 (0.160)
  Neutrophil Count Week 0 | 5.6 (0.062) | 5.1 (0.064)
  Neutrophil Count Week 4: number analyzed (Participants) | 42 | 36
  Neutrophil Count Week 4 | 4.9 (0.046) | 4.9 (0.049)
  Neutrophil Count Week 12: number analyzed (Participants) | 42 | 35
  Neutrophil Count Week 12 | 5.4 (0.053) | 5.2 (0.059)
  Neutrophil Count Week 24: number analyzed (Participants) | 39 | 36
  Neutrophil Count Week 24 | 5.4 (0.059) | 5.0 (0.061)
  Neutrophil Count Week 36: number analyzed (Participants) | 39 | 36
  Neutrophil Count Week 36 | 5.6 (0.056) | 4.9 (0.059)
  Neutrophil Count Week 48: number analyzed (Participants) | 20 | 16
  Neutrophil Count Week 48 | 5.3 (0.079) | 5.5 (0.089)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; White blood cell count; Test type: Superiority; p = 0.736, Mixed Models Analysis — Outcome was log transformed Explanatory variables: treatment arm, number of exacerbations in the 12 months prior to the trial (stratification factor), log BL value, visit time point (categorical) and patient identification (random effect); Geometric mean ratio = 1.01, 95% CI 2-sided [0.95 to 1.07]
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; Eosinophil Count; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Geometric mean ratio = 0.59, 95% CI 2-sided [0.51 to 0.69]
Statistical Analysis 3: Comparison: Anti-ST2 vs Placebo; Neutrophil Count; Test type: Superiority; p = 0.678, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]; Geometric mean ratio = 1.02, 95% CI 2-sided [0.93 to 1.13]

13. Secondary Outcome: Sputum Inflammatory Cell Differentials: Eosinophils
Description: To assess inflammation at exacerbation events. Eosinophils cells will be measured.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Geometric Mean (Standard Error); unit: Percentage of Eosinophils in sputum
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 31 | 34
Percentage of Eosinophils in sputum
  Eosinophil count (%) Week 0 | 1.42 (0.254) | 1.63 (0.242)
  Eosinophil count (%) Week 4: number analyzed (Participants) | 29 | 30
  Eosinophil count (%) Week 4 | 0.43 (0.188) | 1.69 (0.185)
  Eosinophil count (%) Week 12: number analyzed (Participants) | 31 | 24
  Eosinophil count (%) Week 12 | 0.41 (0.168) | 1.67 (0.190)
  Eosinophil count (%) Week 24: number analyzed (Participants) | 24 | 20
  Eosinophil count (%) Week 24 | 0.44 (0.191) | 1.69 (0.209)
  Eosinophil count (%) Week 36: number analyzed (Participants) | 26 | 21
  Eosinophil count (%) Week 36 | 0.47 (0.212) | 1.94 (0.236)
  Eosinophil count (%) Week 48: number analyzed (Participants) | 11 | 10
  Eosinophil count (%) Week 48 | 0.33 (0.232) | 1.24 (0.243)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Eosinophil count; Test type: Superiority; p < 0.001, Mixed Models Analysis — A mixed effect linear model of the log outcome with explanatory variables treatment, number of exacerbations in the 12 months prior to the trial (stratification), visit time point (as categorical variable) and log baseline score as fixed effects; Geometric mean ratio = 0.25, 95% CI 2-sided [0.19 to 0.33]

14. Other Pre Specified Outcome: Non-contrast Thoracic CT Derived Outcomes [Exploratory Outcome]
Description: Quantitative measures of airway geometry and densitometry. Mean lung density expiratory/inspiratory [MLD E/I] (small airway), % wall area [WA] and LA (larger airways) will be measured.
Time Frame: Screening and week 48
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Sputum Mediator Profiling (Biomarkers) [Exploratory Outcome]
Description: Various biomarkers of inflammation will be measured in sputum.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Blood Biomarkers [Exploratory Outcome]
Description: Various biomarkers of inflammation will be measured in blood.
Time Frame: Screening, weeks 4, 12, 24, 36, 48
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Cell Subset Analysis Including But Not Restricted to Exploration of ILC2 Cells [Exploratory Outcome]
Description: ILC2 cells will be analysed using plasma for biomarkers.
Time Frame: Screening, weeks 4, 12, 24, 36, 48
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Urine Biomarkers of Inflammation [Exploratory Outcome]
Description: Various biomarkers of inflammation will be measured in urine.
Time Frame: Screening, weeks 0, 4, 12, 24, 36, 48
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Mediator Profiling (Biomarkers) [Exploratory Outcome]
Description: Mediators of inflammation in blood, sputum and urine will be assessed.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Nasosorption [Exploratory Outcome]
Description: To assess upper airway inflammation. This is a non-invasive method to sample nasal mucosal lining fluid using a synthetic absorptive matrix (SAM) of low protein binding. The SAM is advanced up the lumen of the nasal cavity, and then the outside of the nose is gently pressed to oppose the SAM against the nasal mucosa for 30 seconds.
Time Frame: Screening, Weeks 12, 24, 36, 48
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Nasal Epithelial Sampling [Exploratory Outcome]
Description: To assess airway upper inflammation. Nasal epithelial cells will be sampled from the anterior nares using either a polyester swab or a cytology brush with the standard collection method - cytology brush sampling from beneath the inferior turbinate. This test is optional for participants.
Time Frame: Screening, weeks 12, 24, 36, 48
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Breath Volatile Organic Compound (VOC) Profiling [Exploratory Outcome]
Description: To assess inflammation. PTR-MS, ADVION and ReCIVA will be used to measure gaseous molecules found in the breath that are from inside and outside the lungs. We aim to collect these molecule and analyse them to see if there are any changes in a persons breath that could be linked to the metabolic health, before, during and after taking the drug or placebo.
Time Frame: Screening, Weeks 12, 24, 36, 48
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Microbiomics [Exploratory Outcome]
Description: To assess airway infection and ecology. We will analyse the microbes in patients' lungs using their sputum samples and profile the effect of treatment on these microbes.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Targeted qPCR (Bacteria and Viruses) for Common Airway Pathogens [Exploratory Outcome]
Description: To assess airway infection and ecology. We will analyse the microbes in patients' lungs and profile the effect of treatment on these microbes.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Pharmacogenomics Response Analysis in Subgroups Determined by SNPs for Alleles Associated With the IL33/ST2 Axis. [Exploratory Outcome]
Description: To evaluate the rate of protocol-defined COPD exacerbations through 48 weeks treatment period, patient reported outcomes (PROs), and lung functions, by subgroup outcomes.
Time Frame: Baseline and week 48
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Baseline Blood Eosinophil Count [Subgroup Objective]
Description: To evaluate the efficacy of anti-ST2 versus placebo on the outcome rate of protocol-defined COPD exacerbations through 48 weeks treatment period, patient reported outcomes (PROs) and lung function in subgroups defined by baseline blood eosinophil count.
Time Frame: Screening, weeks 4, 12, 24, 36, 48
Reporting Status: Not Posted

27. Other Pre Specified Outcome: St George's Respiratory Questionnaire for COPD Patients (SGRQ-c) [Subgroup Objective]
Description: as for outcome 26
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Reporting Status: Not Posted

28. Other Pre Specified Outcome: FEV1 [Subgroup Objective]
Description: as for outcome 26
Time Frame: Weeks 0 and 48
Reporting Status: Not Posted

29. Secondary Outcome: Pre and Post Bronchodilator (BD) Spirometry- FEV1 and FVC
Description: To assess lung function. The participant will take a maximum inhalation, release maximum exhalation and then continue to exhale afterwards. They will then be treated with a bronchodilator. The spirometry test is then repeated to determine how much the bronchodilator medication helped with breathing. FEV1 and FVC will be measured.
Time Frame: Week 0 and Week 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 8 | 5
Litres
  Pre BD FEV1 Week 0 | 1.43 (0.43) | 0.94 (0.33)
  Pre BD FEV1 Week 48 | 1.43 (0.49) | 0.86 (0.15)
  Pre BD FVC Week 0 | 2.97 (0.89) | 2.17 (0.34)
  Pre BD FVC Week 48 | 2.88 (0.94) | 2.20 (0.36)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Pre BD FVC (litres): Analysis of covariance (ANCOVA) adjusting for the baseline value; Test type: Superiority; p = 0.362, ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.14 to 0.35]
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; Pre BD FVC (litre):Analysis of covariance (ANCOVA) adjusting for the baseline value; Test type: Superiority; p = 0.713, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.61 to 0.44]

30. Secondary Outcome: Pre and Post Bronchodilator (BD) Spirometry- FEV1 Predicted and FVC Predicted
Description: To assess lung function. The participant will take a maximum inhalation, release maximum exhalation and then continue to exhale afterwards. They will then be treated with a bronchodilator. The spirometry test is then repeated to determine how much the bronchodilator medication helped with breathing. FEV1 % predicted and FVC % predicted will be measured.
Time Frame: Week 0 and Week 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 8 | 5
Percent predicted
  Pre BD FEV1 predicted (%) Week 0 | 55.9 (17.1) | 39.6 (10.4)
  Pre BD FEV1 predicted (%) Week 48 | 56.5 (19.9) | 38.2 (8.3)
  Pre BD predicted FVC (%) Week 0 | 88.5 (16.6) | 75.6 (16.7)
  Pre BD predicted FVC (%) Week 48 | 85.8 (22.8) | 79.2 (28.5)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Pre FEV1 predicted: Analysis of covariance (ANCOVA) adjusting for the baseline value; Test type: Superiority; p = 0.711, ANCOVA; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-8.63 to 12.20]
Statistical Analysis 2: Comparison: Anti-ST2 vs Placebo; Pre BD FVC predicted (%): Analysis of covariance (ANCOVA) adjusting for the baseline value; Test type: Superiority; p = 0.214, ANCOVA; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-27.9 to 7.1]

31. Secondary Outcome: Body Plethysmography ('Body Box') - Residual Volume/Total Lung Capacity Ratio
Description: To assess lung function, i.e. the functional residual capacity of the lungs. The participant sits inside an airtight box, inhales or exhales to a particular volume (usually FRC), and then a shutter drops across their breathing tube. The participant makes respiratory efforts against the closed shutter, causing their chest volume to expand and decompressing the air in their lungs. The increase in their chest volume slightly reduces the box volume (the non-person volume of the box) and thus slightly increases the pressure in the box. Residual Volume/Total Lung Capacity ratio will be calculated. RV/TLC ratio: this is the residual volume (RV) to total lung capacity (TLC). It is calculated as a percentage as follows: RV/TLC ×100.
Time Frame: Week 0 and week 48
Population: Modified ITT (available data)
Measure: Mean (Standard Deviation); unit: percentage (RV of TLC)
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 19 | 16
percentage (RV of TLC)
  Residual Volume/Total Lung Capacity ratio (%) Week 0 | 59.8 (9.5) | 61.3 (11.5)
  Residual Volume/Total Lung Capacity ratio (%) Week 48 | 61.1 (11.2) | 65.2 (9.7)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Residual Volume/Total Lung Capacity ratio; Test type: Superiority; p = 0.201, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-7.53 to 1.65]

32. Secondary Outcome: Sputum Inflammatory Cell Differentials: Macrophages
Description: To assess inflammation at exacerbation events. Sputum inflammatory cell differentials: Macrophages
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Geometric Mean (Standard Error); unit: Percentage of Macrophage in sputum
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 31 | 34
Percentage of Macrophage in sputum
  Macrophage count in sputum (%) Week 0 | 8.9 (0.205) | 9.6 (0.196)
  Macrophage count in sputum (%) Week 4: number analyzed (Participants) | 29 | 30
  Macrophage count in sputum (%) Week 4 | 8.6 (0.211) | 11.0 (0.208)
  Macrophage count in sputum (%) Week 12: number analyzed (Participants) | 31 | 24
  Macrophage count in sputum (%) Week 12 | 9.0 (0.190) | 9.8 (0.216)
  Macrophage count in sputum (%) Week 24: number analyzed (Participants) | 24 | 20
  Macrophage count in sputum (%) Week 24 | 9.2 (0.222) | 12.3 (0.244)
  Macrophage count in sputum (%) Week 36: number analyzed (Participants) | 26 | 21
  Macrophage count in sputum (%) Week 36 | 8.1 (0.213) | 9.7 (0.237)
  Macrophage count in sputum (%) Week 48: number analyzed (Participants) | 11 | 10
  Macrophage count in sputum (%) Week 48 | 6.9 (0.286) | 11.4 (0.300)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Macrophage count; Test type: Superiority; p = 0.114, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]; Geometric mean ratio = 0.75, 95% CI 2-sided [0.52 to 1.07]

33. Secondary Outcome: Sputum Inflammatory Cell Differentials: Epithelium
Description: To assess inflammation at exacerbation events. Epithelium cells will be measured.
Time Frame: Weeks 0, 4, 12, 24, 36, 48
Population: Modified ITT (available data)
Measure: Geometric Mean (Standard Error); unit: Percentage of Epithelium in sputum
Arm/Group | Anti-ST2 | Placebo
Number analyzed (Participants) | 31 | 34
Percentage of Epithelium in sputum
  Epithelium count (%) Week 0 | 1.51 (0.255) | 1.59 (0.243)
  Epithelium count (%) Week 4: number analyzed (Participants) | 29 | 30
  Epithelium count (%) Week 4 | 1.34 (0.257) | 2.06 (0.253)
  Epithelium count (%) Week 12: number analyzed (Participants) | 31 | 24
  Epithelium count (%) Week 12 | 1.14 (0.243) | 1.91 (0.276)
  Epithelium count (%) Week 24: number analyzed (Participants) | 24 | 20
  Epithelium count (%) Week 24 | 1.56 (0.284) | 1.44 (0.311)
  Epithelium count (%) Week 36: number analyzed (Participants) | 26 | 21
  Epithelium count (%) Week 36 | 1.03 (0.266) | 1.26 (0.296)
  Epithelium count (%) Week 48: number analyzed (Participants) | 11 | 10
  Epithelium count (%) Week 48 | 1.56 (0.435) | 1.21 (0.456)
Statistical Analysis 1: Comparison: Anti-ST2 vs Placebo; Epithelium count; Test type: Superiority; p = 0.215, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]; Geometric mean ratio = 0.79, 95% CI 2-sided [0.54 to 1.15]

ADVERSE EVENTS:
Time Frame: Adverse event data occurring from the point of randomisation until the final trial visit following follow-up (or 100 days post cessation of trial treatment (if discontinued early), were recorded throughout the 48 week treatment period and 12 week post-trial follow-up.
Arm/Group | Anti-ST2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 2/39
Serious Adverse Events (participants affected / at risk) | 12/42 | 16/39
Other Adverse Events (participants affected / at risk) | 34/42 | 28/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-ST2 (N=42) | Placebo (N=39)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adenoma of the bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood transfusion (anaemia) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest infection/infective exacerbation of bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Clinical diagnosis of lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Descending aorta thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Elective surgery (transurethral resection of the prostate) (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymo-orchitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Flu-like illness (viral infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fractured neck of femur (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hospital acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Infective exacerbation of bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Left scaphoid fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oesophageal cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonia and type 2 respiratory failure (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Resection of prostate (Renal and urinary disorders) | 1 (1) | 0 (0)
Right pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right thrombosed popliteal aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suspected UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncopal episode (Cardiac disorders) | 0 (0) | 1 (1)
Type 2 respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-ST2 (N=42) | Placebo (N=39)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Chest pain (General disorders) | 5 (5) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 10 (20) | 5 (9)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Lethargy (General disorders) | 2 (2) | 2 (2)
Malaise (General disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (11) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 3 (5) | 4 (6)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (2)

LIMITATIONS AND CAVEATS:
* Small sample size (n=81) at a single site, therefore not powered to detect a reduction in exacerbation frequency that was observed.
* Participants were required to have had a minimum of 2 exacerbations in the previous 12 months, so the findings are not representative for a wider clinical population.
* In response to COVID-19, collection of secondary/exploratory outcomes were reduced, with spirometry and sputum induction discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT03615040/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03615040/SAP_001.pdf
  • Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03615040/ICF_002.pdf